CLINICAL TRIAL: NCT00151307
Title: The Effects of Monitoring and Maintaining Cerebral Oxygen Saturation on Neuropsychological Outcomes in Patients Undergoing Cardiac Surgery
Brief Title: Effects of Cerebral Oxygen Saturation on Neuropsychological Outcomes
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Could not recruit any more people.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0599-691
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Cardiovascular Diseases; Postoperative Complications
Keywords: Heart surgery; Cerebral oxygen saturation; Neuropsychological function
MeSH Terms: conditions — Cardiovascular Diseases; Postoperative Complications

INTERVENTIONS:
Device: INVOS cerebral oximeter

SUMMARY:
The purpose of this study is to evaluate the effects of maintaining adequate cerebral oxygen saturation (over 40%) on patients undergoing cardiac surgery. Effects on neuropsychological outcome, length of ICU stay, and length of hospital stay will be measured.

DETAILED DESCRIPTION:
Central nervous system dysfunction is a major cause of morbidity after cardiac surgery. This study seeks to evaluate the effects of cerebral oxygen saturation on the neuropsychological outcome of cardiac surgery patients. Currently, monitoring of cerebral oxygen saturation levels is not part of routine and standard practice.

Subjects will be assigned to a control and intervention group. Anesthesia and surgery will be performed as per usual standards of care. Patients in both groups will be monitored with an oxygen sensor placed over the forehead. The data will be recorded continuously on a floppy disk. The control group will be treated according to current standard of care; the readings of brain oxygen saturation will not be visible to the clinician. In the intervention group, the reading of brain oxygen saturation will be monitored by the anesthesiologist throughout surgery. Interventions will be performed to maintain cerebral oxygen saturations above 40%. Neuropsychological tests will be completed pre-operatively and at two time points post-operatively. The tests used are the ASEM (antisaccadic eye movement) and the MMSE (mini-mental state examination).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Elective cardiac surgery with cardiopulmonary bypass
* Coronary artery disease or valvular heart disease or combination of both
* Ability and willingness to give informed consent

Exclusion Criteria:

* Pediatric patients
* Emergency surgery
* Unable to understand English
* Allergic to tape used to attach oxygen sensor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2001-02; Study Completion 2007-04

PRIMARY OUTCOMES:
Neuropsychological Outcome
Tests:
Anti-saccadic eye movement
Mini-mental state examination
Neurological testing
Completed pre-operatively, 3-4 days post-op, 2-3 months post-op

SECONDARY OUTCOMES:
ICU & Hospital length of stay
Morbidity (complications post-op)
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Fun-Sun Yao, M.D., Principal Investigator — Anesthesiology; Weill Medical College of Cornell University, New York Presbyterian Hospital
Locations (1):
- New York Presbyterian Hospital, Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Yao FS, Tseng CC, Ho CY, Levin SK, Illner P. Cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Oct;18(5):552-8. doi: 10.1053/j.jvca.2004.07.007. PMID 15578464